CLINICAL TRIAL: NCT03137862
Title: A Prospective, Double Blind, Placebo-controlled Trial to Evaluate Efficacy and Safety of a "Gluten Friendly" Bread in Population With Celiac Disease
Brief Title: "Gluten Friendly" Treatment in Celiac Disease
Acronym: GLUFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: University of Foggia (Other)
Responsible Party: Principal Investigator, Angelo Andriulli, Chief of Gastroenterology and Digestive Endoscopy CSDSofferenza, Casa Sollievo della Sofferenza IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NCT64/CE
Record Dates: First submitted 2017-04-10; First posted 2017-05-03 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Food Intolerance; Celiac Disease
MeSH Terms: conditions — Food Intolerance; Celiac Disease

STUDY DESIGN:
Intervention Model Description: double blind prospective study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A comparator (Placebo Comparator): Arm A: patients will maintain a commercially available gluten free diet and receive bread containing 3 gr of cornstarch daily for 12 weeks; these patients will serve as controls.
  Interventions: Other: Gluten free bread
- Arm B (Experimental): Dietary supplement: patients will be have to continue the gluten free diet supplemented with 3 gr of "gluten friendly" bread daily for 12 weeks.
  Interventions: Other: Gluten free bread; Dietary Supplement: Gluten friendly bread 3g/day
- Arm C (Experimental): Dietary supplement: patients will be have to continue the gluten free diet supplemented with 6 gr of "gluten friendly" bread daily for 12 weeks
  Interventions: Dietary Supplement: Gluten friendly bread 6g/day

INTERVENTIONS:
Other: Gluten free bread — patients will receive bread containing 3 g of cornstarch daily for 12 weeks; these patients will serve as controls
  Arms: Arm A comparator; Arm B
Dietary Supplement: Gluten friendly bread 3g/day — patients will have to continue the GFD supplemented with 3 gr of "gluten friendly" bread daily for 12 weeks
  Arms: Arm B
Dietary Supplement: Gluten friendly bread 6g/day — patients will have to continue the GFD supplemented with 6 gr of "gluten friendly" bread daily for 12 weeks
  Arms: Arm C

SUMMARY:
A PROSPECTIVE, double blind, placebo-controlled trial

DETAILED DESCRIPTION:
Background: Gluten ingestion leads to small intestinal mucosal injury in patients with celiac disease (CD), necessitating rigid, life-long exclusion of gluten from diet. Current therapies based on gluten-free dietary regimes, are also impairing social life, increased expenses for gluten free products, personal dissatisfaction and frustration. In addition, gluten-free products often have a low content of vitamins, such as vitamins B, ions such as calcium, iron, zinc and magnesium, as well of fibres. An alternative to the exclusion of gluten from diet may be the detoxification of gluten without affecting the technological performance of the flour and dough. Recently, we succeeded in developing a new and innovative method to detoxify gluten proteins from cereal grains: the modified stuff was capable to retain nutritional and technological properties of wheat proteins, and proved to be safe to celiac and gluten-sensitive patients. This innovation is usually referred to as "gluten friendly".

Objective: To establish the efficacy and safety of a prolonged exposure to the "Gluten Friendly trademark (™)" bread in patients with celiac disease.

Design: A prospective, double-blind, placebo-controlled, randomized trial to be conducted on adults with biopsy-proven CD who were being treated with a gluten-free diet (GFD) for >2 years. Before enrollment, consenting patients will have to sign an informed consent form with full details of the aims of the study, and an explanation of the experimental procedures of the study. At the baseline evaluation (t 0 ), patients will undergo a clinical examination, an upper gastrointestinal endoscopy for the histologic evaluation of the duodenal mucosa, and a blood drawing for routine chemistry and anti-transglutaminase (ATGA) and anti-endomysium (EMA) antibodies checking. Eligible to be enrolled into the study will be patients with undetectable ATGA and EMA antibodies. They will be randomly assigned to one of three experimental regimens:

1. the control arm: patients will maintain a commercially available GFD and receive bread containing 3 gr of cornstarch daily for 12 weeks; these patients will serve as controls (Group A)
2. the innovative arm 1: patients will be have to continue the GFD supplemented with 3 gr of "gluten friendly"™ bread daily for 12 weeks (Group B)
3. the innovative arm 2: patients will be have to continue the GFD supplemented with 6 gr of "gluten friendly"™ bread daily for 12 weeks (group C).

All patients will be provided with a diary card to monitor their adherence to the assigned treatments and to register their acceptance of the experimental breads. Either patients and attending physicians will maintain blindness about the treatment assignment throughout t the study period.

At the end of the 2nd and 4th treatment week, patients will be monitored for ATGA and EMA antibodies, and those with positive results will undergo a repeat endoscopy for checking the integrity of the duodenal mucosa: in the event of any deterioration of histology, patients will patients will be considered as treatment failures. Patients with negative serology will be kept on treatment for the scheduled 12 weeks. At 12th week, patients will have to return for a clinical examination, a repeat blood drawing for ATGA, anti-EMA, anti-gliadin (AGA both IgG and IgA) antibodies checking, immunoglobulin G (IgG), immunoglobulin A (IgA), routine chemistry, complete hematology work up including serum iron, phosphorus, folate, and vitamin D3 measurements. In addition, a new, repeat endoscopy will be scheduled for all enrolled patients with the intent to acquire information on the histologic status of the duodenal mucosa, the the principal outcome of this investigation. After the completion of the 12 weeks study period, all patients will be invited to enter in an open study in which the addition of the "Gluten Friendly ™" bread to their GFD diet will be administered for a very long period of time, likely 6 or 12 months. This section of the study will be run on a voluntary basis and will serve to gain information about safety of the modified gluten in the long run.

ELIGIBILITY:
Inclusion Criteria:

* celiac patients with positive antitransglutaminase and histology compatible with celiac disease

Exclusion Criteria:

* positive antitransglutaminase at enrollment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-04-02 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Measure of small bowel mucosal density and evaluation of the serologic markers of celiac disease | Three months after of treatment
  Endoscopy evaluation of duodenum and determination of anti-tTG2-IgA, EMA and AGA antibodies levels

CONTACTS AND LOCATIONS:
Locations (1):
- Angelo Andriulli, San Giovanni Rotondo, FG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andriulli A, Bevilacqua A, Palmieri O, Latiano A, Fontana R, Gioffreda D, Castellana S, Mazza T, Panza A, Menzaghi C, Grandone E, di Mauro L, Decina I, Tricarico M, Musaico D, Maki M, Isola J, Popp A, Taavela J, Petruzzi L, Sinigaglia M, Rosaria Corbo M, Lamacchia C. Healthy and pro-inflammatory gut ecology plays a crucial role in the digestion and tolerance of a novel Gluten Friendly bread in celiac subjects: a randomized, double blind, placebo control in vivo study. Food Funct. 2022 Feb 7;13(3):1299-1315. doi: 10.1039/d1fo00490e. PMID 35029612